CLINICAL TRIAL: NCT02113124
Title: Association of Amino Acid Prevalence and Chronic Brain Injury
Status: Completed | Type: Observational
Sponsor: Brent Masel (Other)
Collaborators: The Moody Foundation (Other)
Responsible Party: Sponsor-Investigator, Brent Masel, Brent Masel, M.D., The Transitional Learning Center, Galveston, TX
Organization: The Transitional Learning Center, Galveston, TX (Other)
Other Study IDs: TLC IRB #200
Record Dates: First submitted 2014-04-08; First posted 2014-04-14 (Estimated); Results first posted 2015-11-17 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Traumatic Brain Injury
Keywords: Chronic Brain Injury; Traumatic brain injury (TBI); Amino Acids; Microbiome
MeSH Terms: conditions — Brain Injury, Chronic; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood, oral tissue swab, fecal matter
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic brain injury: Individuals in this group have suffered a brain injury more than 2 years prior to study. Ages range from 21 to 70.
- Uninjured control: This group of individuals have no history of brain injury. Ages range between 21 and 70.

SUMMARY:
Years after a suffering a brain injury, individuals remain in a physically and cognitively impaired state. The investigators believe that the concentrations of amino acids in the blood are chronically altered and yield negative effects on the individuals health. Preliminary data has shown significantly lower concentrations of amino acids in serum samples from the TBI population, these diminished levels of amino acids may be due to changes in the microbiome. Understanding these changes will help guide rehabilitative services for this population. Individuals with a chronic brain injury will donate samples of blood, oral tissue, and fecal matter to be compared to that of non-injured individuals. Genetic information from the hosts will be striped and discarded; participant's genetic information will not be retained. To better understand changes in the microbiome, any history of antibiotics and probiotics will be assessed.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the levels of Amino Acids in adult individuals with chronic (> 2 years) traumatic brain injury (TBI) when compared to a non-brain injured cohort population.

Preliminary data from an assay of amino acids in individuals with chronic TBI compared to an assay of individuals without a TBI revealed significantly lower concentrations of amino acids within the TBI group.

The composition and structure of the oral and fecal microbiome will be determined by 16S rDNA sequencing. Taxonomic and community structure profiles will be treated as outcome variables and modeled together with the participant's plasma amino acid concentration, years post-injury, age, sex and other variables to determine correlations. These correlations may improve our understanding of the diminished amino acid metabolism within the chronic TBI population.

The endpoint will identify the microbiome structure and composition by 16S rRNA gene sequencing within the TBI and healthy participants and to assess the participant's amino acid concentrations and other participant demographics and phenotypic characteristics (years post-injury, age, sex). This comparison may improve our understanding of the diminished amino acid metabolism within the chronic TBI population.

ELIGIBILITY:
Inclusion Criteria:

* Willing to donate 10 ml of blood
* Willing to donate oral tissue sample
* Willing to donate fecal sample

Exclusion Criteria:

* (for brain injured group) have a chronic (greater than two years) traumatic brain injury.
* Unable to provide to give voluntary informed consent

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals in the chronic brain injured group are recruited from traumatic brain injury rehabilitation facilities. These facilities include Tideway in Galveston, Texas, Centre for Neuro Skills in Bakersfield, CA, and Centre for Neuro Skills in Dallas, TX. The cohorts for this study will be recruited from the communities surrounding the rehabilitation facilities.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent E Masel, MD, Principal Investigator — Transitional Learning Center
Locations (3):
- United States (3):
  - Centre for Neuro Skills, Bakersfield, California
  - Centre for Neuro Skills, Dallas, Texas
  - Transitional Learning Center, Galveston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic Brain Injury: Individuals in this group have suffered a brain injury more than 2 years prior to study. Ages range from 35 to 70.
- Uninjured Control: This group of individuals have no history of brain injury. Ages range between 35 and 70.
Period: Overall Study
Arm/Group | Chronic Brain Injury | Uninjured Control
Started | 18 | 25
Completed | 17 | 24
Not Completed | 1 | 1
Not completed — Unable to retrieve blood sample | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Brain Injury | Uninjured Control | Total
Number analyzed (Participants) | 17 | 24 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (10) | 45 (15) | 46 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 8
  Male | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Concentrations of Essential Amino Acid at 1.5 Hours After Eating
Description: 5 ml of blood will be acquired following a 8-hour fasting period to determine baseline concentrations of amino acids. A meal will then be provided and another blood sample will be acquired 90 minutes after completing the meal to examine the change in amino acid concentration. These samples will be used to determine the levels of each essential amino acid present.
Time Frame: Samples collected on day 1 following 8 hour fasting period and again 90 minutes after eating a predetermined meal
Measure: Mean (Standard Error); unit: µM
Arm/Group | Chronic Brain Injury | Uninjured Control
Number analyzed (Participants) | 17 | 24
µM
  Branched Chain Amino Acids | 487.28 (22.94) | 553.70 (38.26)
  Essential Amino Acids | 1224.19 (27.50) | 1339.54 (73.17)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected on day 1 immediately following each blood draw, for up to 8 hours.
Arm/Group | Chronic Brain Injury | Uninjured Control
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/25
Other Adverse Events (participants affected / at risk) | 0/18 | 0/25

LIMITATIONS AND CAVEATS:
No limitations reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes